CLINICAL TRIAL: NCT05332418
Title: EFFECT OF ELECTROMAGNETIC FIELD THERAPY ON NECK PAIN AND PROPRIOCEPTION IN CERVICAL RADICULOPATHY PATIENTS
Brief Title: ELECTROMAGNETIC FIELD ON NECK PAIN AND PROPRIOCEPTION IN CERVICAL RADICULOPATHY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Lama Saad El-Din Mahmoud, Lecturer of physical therapy, Department of Neuromuscular disorders and its surgery, faculty of physical therapy, october 6 univerisity, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T. REC/012/003565
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Intervention Model Description: the control group which received the selected exercise program and the study group received the same exercise training program in addition to electromagnetic field therapy, three times per week for four weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): the study group received the same exercise training program in addition to electromagnetic field therapy, three times per week for four weeks
  Interventions: Other: selected exercise program; Device: Electromagenetic Field therapy
- control group (Experimental): the control group which received the selected exercise program
  Interventions: Other: selected exercise program

INTERVENTIONS:
Other: selected exercise program — therapeutic ultrasound, Static neck exercise, Educational postural correction, and Home neck exercise program for patient
Device: Electromagenetic Field therapy — Magnetotherapy application the device will be adjusted around the neck and shoulder area at low frequency (50 Hz), with intensity of 2.5 MT, field shape and applicator type rectangular csl60/csp60) , and the application time (10 minutes)
  Arms: study group

SUMMARY:
PURPOSE:

to investigate effect of electromagnetic field therapy on neck pain and proprioception in cervical radiculopathy patients

BACKGROUND: Cervical radiculopathy is a clinical condition resulting from compression of cervical nerve roots Pulsed electromagnetic field (PEMF) therapy is an easy, non-invasive, safe, and relatively new treatment method that is used with growing interest in physical and rehabilitation medicine. Historically, the benefits from magnetotherapy have been reported for patients with musculoskeletal and neurological disorders

DETAILED DESCRIPTION:
Thirty four patients with cervical radiculopathy The patients will randomly be divided into two equal groups; the control group which received the selected exercise program and the study group received the same exercise training program in addition to electromagnetic field therapy, three times per week for four weeks. The evaluation methods by Visual analogue scale for pain (VAS-P), cervical joint position error test (JPET), Neck disability index , and Cervical range of motion (CROM) goniometer device measurements

ELIGIBILITY:
Inclusion Criteria:

1. Age ranging from 30:45
2. Cervical radiculopathy due to disc prolapse (C5-C6) (C6-C7) mild to moderate or disc prolapse according to magnetic resonance image (MRI).
3. With mild to moderate cervical disability according to neck disability index
4. Body mass index (18.5 to 29.9) Kg/m2.

Exclusion Criteria:

1. Cervical myelopathy.
2. Patients with previous cervical surgery.
3. Inflammatory diseases such as rheumatoid arthritis or ankylosing spondylitis
4. Any other musculoskeletal disorders of the spine or upper extremity.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale for pain (VAS-P) | 4 weeks
  is a method for measuring the intensity of pain on a horizontal straight line of fixed length (10 cm), as the left end of the line showed the greatest pain score & the right end showed the least pain scores, then the patient was asked to put a mark, on the line according to his/her pain sensation, with a higher score representing the higher level of pain
cervical proprioception using cervical joint position error test (JPET) | 4 weeks
  * The subject will be instructed to perform an active head rotation to one side, after which returns back to the neutral or starting head position.
  * The test will be performed in a 3 trials in each direction: right, left rotations , extension and flexion.
Neck disability index | 4 weeks
  includes 10 items as follows: Pain Intensity, Personal Care, Lifting, Reading, Headaches, Concentration, Work, Driving, Sleeping, and Recreation, with a score (0:5) for every point. The maximum score is 50, with the interpretation scoring (no disability = 0: 4, mild disability 5:14, moderate disability 15:24, severe disability 25: 34 and complete disability above 34
Cervical range of motion (CROM) goniometer device | 4 weeks
  The CROM is an inclinometers system with a gravitational reference that is suitable for evaluating the active cervical spine movements in different direction

CONTACTS AND LOCATIONS:
Locations (1):
- Lama Saad El-Din Mahmoud, Al Jīzah, Select State, Egypt